CLINICAL TRIAL: NCT03945747
Title: MEtabolic and Renal Effects of AutoMAted Insulin Delivery Systems in Youth With Type 1 Diabetes Mellitus (MERMAID-T1D)
Brief Title: MEtabolic and Renal Effects of AutoMAted Insulin Delivery Systems in Youth With Type 1 Diabetes Mellitus
Acronym: MERMAID-T1D
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Colorado Clinical & Translational Sciences Institute (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-1558; UL1TR002535 (NIH); 5T32DK063687-15 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Type1 Diabetes Mellitus; Diabetes Mellitus, Type 1; Autoimmune Diabetes; Juvenile Diabetes; Diabetes Mellitus Complication; Diabetic Nephropathies; Metabolic Disease; Diabetic Kidney Disease
Keywords: Automated insulin delivery systems; Insulin sensitivity; Cardiometabolic function; Renal function
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Complications; Diabetic Nephropathies; Metabolic Diseases; Insulin Resistance | interventions — Blood Specimen Collection; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Individuals continue current treatment regimen with either standard insulin pump therapy or multiple daily insulin injections for the duration of the study.
  Interventions: Diagnostic Test: Blood draw; Diagnostic Test: Urine sample collection; Diagnostic Test: DXA scan
- Hybrid closed-loop artificial pancreas system group: Individuals transition from either standard insulin pump therapy or multiple daily injections to a hybrid closed-loop system at the beginning of the study after initial labs and imaging studies are completed.
  Interventions: Diagnostic Test: Blood draw; Diagnostic Test: Urine sample collection; Diagnostic Test: DXA scan
- Predictive low glucose suspend system group: Individuals transition from either standard insulin pump therapy or multiple daily injections to a predictive low glucose suspend system at the beginning of the study after initial labs and imaging studies are completed.
  Interventions: Diagnostic Test: Blood draw; Diagnostic Test: Urine sample collection; Diagnostic Test: DXA scan

INTERVENTIONS:
Diagnostic Test: Blood draw — Participants will undergo a blood collection for hemoglobin A1c, adiponectin, total cholesterol, LDL, HDL, triglycerides, and c-peptide at baseline and follow up in 3-6 months.
Diagnostic Test: Urine sample collection — Participants will undergo urine sample collection for urine microalbumin and urine creatinine at baseline and follow up in 3-6 months.
Diagnostic Test: DXA scan — Participants will undergo a DXA scan for lean and fat mass measurements at baseline and follow up in 3-6 months.

SUMMARY:
In type 1 diabetes (T1DM), automated insulin delivery (AID) systems such as the hybrid closed loop artificial pancreas (HCL AP) combine the use of an insulin pump, continuous blood sugar monitor, and control algorithm to adjust background insulin delivery to improve time in target blood sugar range. Systems such as the predictive low glucose suspend system (PLGS) pause insulin delivery to try and reduce low blood sugars. We aim to complete a pilot study involving recruitment of youth ages 7 to 18 years from the following groups with type 1 diabetes: control participants consisting of youth on either multiple daily insulin injections or conventional insulin pump therapy that plan to continue with their current treatment modality, youth being transitioned to the HCL AP system, and youth being transitioned to the PLGS system. Individuals will be recruited into each of the aforementioned study groups based on their own expressed desire to either continue on MDI/standard insulin pump therapy or transition to either the HCL AP or PLGS systems. The decision to either continue with current therapy or transition therapy will remain entirely up to the participant and their family and will be based on personal preference and insurance coverage for that individual. We will not be randomizing the participants to any given treatment group during this study but rather will be recruiting based on the participant's decision. We would like to complete a physical exam with pubertal staging, collect blood and urine samples to evaluate cardiometabolic and renal markers, and complete a DXA scan to evaluate total lean and fat mass. After 3-6 months of either continuation of current treatment with either multiple daily insulin injections or conventional insulin pump therapy or transitioning to the HCL AP or PLGS systems, we would like to repeat the previously described blood, urine, and imaging tests for comparison. We are interested in examining the impact of the HCL AP and PLGS systems on maintaining blood sugars in target range, insulin sensitivity, and markers of cardiometabolic and renal function. We hypothesize that pauses in insulin delivery, as seen in the setting of automated insulin delivery systems, will result in improvements in insulin sensitivity, cardiometabolic markers, and renal function markers.

DETAILED DESCRIPTION:
Background: Over 1.25 million Americans have type 1 diabetes mellitus (T1DM), significantly increasing the risk of early death from cardio-renal disease. Per the American Diabetes Association, only 14% of children with T1DM meet glycemic targets [Wood et al. Diabetes Care 2013; 36:2035-37]. This is a severe and pervasive problem, as a child diagnosed with T1DM today is expected to live up to 17 years less than non-diabetic peers. It is established that time outside of goal glycemic target range increases the likelihood of developing micro- and macro-vascular diabetic complications including diabetic kidney disease (DKD) and cardiovascular disease (CVD). However, metabolic risk factors beyond glycemic control including insulin resistance and obesity are also increasingly recognized to contribute to the increased risk of DKD and CVD. Automated insulin delivery (AID) systems such as the hybrid closed loop artificial pancreas (HCL AP) combine use of an insulin pump, continuous glucose monitor (CGM), and a control algorithm to adjust background insulin delivery to improve time in target range. AID systems such as the predictive low glucose suspend (PLGS) system pause insulin delivery to try to reduce hypoglycemia. AID systems are now seeing markedly increased commercial use; however, the long-term effects on insulin sensitivity, body mass index (BMI), cardio-metabolic markers, and kidney function have not yet been studied. Preliminary basic science research suggests that periods of rest from insulin exposure provided by AID systems may have positive effects on DKD and CVD risk. In this proposal we intend to investigate the gap in knowledge between glycemic changes seen with AID systems and the impact on markers of long-term complications.

Specific Aims and Hypotheses:

Specific Aim 1: To examine the effects of the AID systems on glycemic control and insulin sensitivity as compared to traditional insulin pumps and multiple daily injections in youth with T1DM Hypothesis 1.1: Treatment with the AID systems improves glycemic control in youth with T1DM Hypothesis 1.2: Treatment with the AID systems increases insulin sensitivity and decreases insulin requirement in youth with T1DM

Specific Aim 2: To examine the effects of the AID systems on kidney function and metabolic markers as compared to traditional insulin pumps and multiple daily injections in youth with T1DM Hypothesis 2.1: Treatment with the AID systems improves metabolic markers in youth with T1DM Hypothesis 2.2: Treatment with the AID systems improves kidney function in youth with T1DM

Design: This study is a pilot study aimed at recruiting youth ages 7 to 18 years from the following 3 groups with T1DM: control participants on either multiple daily injections or conventional pump therapy, youth being transitioned to a HCL AP system, and youth being transitioned to a PLGS system. Exclusion criteria include non-T1DM, non-insulin blood glucose altering medications, pregnancy, breastfeeding, or a ketogenic diet. We plan to complete a physical exam with pubertal staging, collect information on recent insulin usage and dosages, fasting serum and urine samples, and a DXA scan before the participant transitions to either a HCL AP or a PLGS system, if applicable. Following 3-6 months of treatment we will then collect the identical data as at baseline. Outcome measures include CGM data, total daily insulin dose, time suspended from insulin delivery, height, weight, BMI, waist circumference, hip circumference, blood pressure, HbA1c, c-peptide, total cholesterol, HDL, LDL, triglycerides, adiponectin, and DXA scan to evaluate cardio-metabolic markers and calculate insulin sensitivity, as well as serum creatinine, cystatin c, copeptin, and urine microalbumin to evaluate kidney health and calculate GFR by Zappitelli and FAS equations.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-18 years
* Type 1 diabetes with at least two of the following criteria: diabetes-associated antibody-positivity, rapid conversion to insulin requirement after diagnosis, absent c-peptide, or DKA at diagnosis
* Currently receiving insulin therapy by multiple daily injections or standard insulin pump therapy

Exclusion Criteria:

* Non-type 1 diabetes mellitus
* Pregnant or breastfeeding
* Receiving treatment with non-insulin glucose-altering medications including oral anti-hyperglycemic medications, steroids, or antipsychotics
* Following a ketogenic diet

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals aged 7-18 years with known type 1 diabetes mellitus who are either planning to continue with standard insulin pump or multiple daily insulin injection therapy OR planning to transition to an automated insulin delivery system such as the hybrid closed-loop artificial pancreas system or the predictive low glucose suspend system.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in estimated insulin sensitivity | 3-6 months
  Estimated by calculating the eIS, Pittsburgh eGDR, and SEARCH IS equations

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (GFR) | 3-6 months
  Estimated by calculating the Zappitelli (CysCrEq) and eGFR-FAS (using serum creatinine) equations
Change in body mass index (BMI) | 3-6 months
  Measured by evaluations of height and weight
Change in lipid profile | 3-6 months
  Measured by fasting blood draw for total cholesterol, LDL, HDL, and triglycerides
Change in c-peptide | 3-6 months
  Measured by fasting blood draw for c-peptide level
Change in DXA scan | 3-6 months
  Evaluation of lean and fat mass by DXA scan

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided